CLINICAL TRIAL: NCT07327892
Title: Comparison of Pericapsular Nerve Group (PENG) Block, PENG Block Plus Periarticular Injection, and Periarticular Injection Alone for Postoperative Pain Management in Older Adults Undergoing Hip Surgery: A Randomized Controlled Trial
Brief Title: PENG Block vs PENG Plus Periarticular Injection vs Periarticular Injection in Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17/2025
Record Dates: First submitted 2025-12-28; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Hip Osteoarthritis; Arthropathy of Hip
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PENG Block (Active Comparator): Participants will receive an ultrasound-guided pericapsular nerve group (PENG) block administered as a single perineural injection prior to surgery, using a standardized technique.
  Interventions: Procedure: Pericapsular Nerve Group (PENG) Block
- PENG Block Plus Periarticular Injection (PAI) (Experimental): Participants will receive an ultrasound-guided PENG block (single perineural injection prior to surgery) plus a periarticular injection administered intraoperatively by the surgeon according to a standardized protocol.
  Interventions: Procedure: Pericapsular Nerve Group (PENG) Block; Procedure: Periarticular Injection (PAI)
- Periarticular Injection (PAI) Alone (Active Comparator): Participants will receive a periarticular injection administered intraoperatively by the surgeon according to a standardized protocol, without a PENG block.
  Interventions: Procedure: Periarticular Injection (PAI)

INTERVENTIONS:
Procedure: Pericapsular Nerve Group (PENG) Block — Ultrasound-guided regional anesthesia technique targeting sensory innervation of the anterior hip capsule, performed as a single injection prior to surgery using a standardized protocol.
  Other Names: Ultrasound-guided PENG block
  Arms: PENG Block; PENG Block Plus Periarticular Injection (PAI)
Procedure: Periarticular Injection (PAI) — Intraoperative periarticular injection performed by the surgeon according to a standardized institutional protocol as part of postoperative pain management.
  Other Names: Local infiltration analgesia; periarticular local anesthetic injection
  Arms: PENG Block Plus Periarticular Injection (PAI); Periarticular Injection (PAI) Alone

SUMMARY:
Pain after hip surgery is common in older adults and may limit early mobilization, increase the need for opioid medications, and contribute to complications such as delirium, nausea, or prolonged hospital stay. Effective postoperative pain management that preserves muscle strength and supports early rehabilitation is especially important in this population.

Several analgesic strategies are currently used after hip surgery. Periarticular injection (PAI), administered by the surgeon during the procedure, is commonly used as part of standard care. The pericapsular nerve group (PENG) block is a newer ultrasound-guided regional anesthesia technique that targets the sensory nerves of the hip joint while sparing motor function. It may provide effective pain relief and facilitate early mobilization. However, it is unclear whether PENG block alone is superior to periarticular injection, and whether combining both techniques provides additional benefit.

The aim of this randomized controlled clinical study is to compare three postoperative analgesic strategies in older adults undergoing hip surgery: PENG block alone, PENG block combined with periarticular injection, and periarticular injection alone. Participants will be randomly assigned to one of three study groups.

The primary hypothesis is that regional anesthesia with a PENG block, either alone or combined with periarticular injection, will provide superior postoperative pain control compared with periarticular injection alone. A secondary hypothesis is that the combination of PENG block and periarticular injection will offer additional analgesic benefit compared with PENG block alone.

Outcomes assessed in this study will include postoperative pain intensity, need for additional pain medications, time to first mobilization, and the occurrence of adverse events relevant to older adults, such as hypotension, excessive sedation, or postoperative delirium.

The results of this study may help determine the most effective and practical analgesic strategy for hip surgery in older adults and support evidence-based optimization of postoperative pain management.

DETAILED DESCRIPTION:
Postoperative pain following hip surgery is a major clinical challenge in older adults and is associated with delayed mobilization, increased opioid consumption, higher risk of delirium, and prolonged hospitalization. Analgesic strategies that provide effective pain relief while preserving motor function are particularly important to support early rehabilitation and reduce postoperative complications in this vulnerable population.

Periarticular injection (PAI), administered intraoperatively by the surgeon, is widely used as part of multimodal analgesia after hip surgery and is considered standard practice in many institutions. The pericapsular nerve group (PENG) block is a relatively new ultrasound-guided regional anesthesia technique designed to selectively block the sensory innervation of the anterior hip capsule while sparing motor nerves. Early clinical data suggest that the PENG block may improve postoperative analgesia and facilitate early mobilization; however, its comparative effectiveness relative to periarticular injection, as well as the potential benefit of combining both techniques, remains insufficiently studied.

This study is designed as a prospective, randomized, controlled, three-arm clinical trial comparing different postoperative analgesic strategies in older adults undergoing hip surgery. Eligible participants will be randomly assigned to one of three groups:

1. PENG block alone,
2. PENG block combined with periarticular injection, or
3. periarticular injection alone. The PENG block will be performed under ultrasound guidance by an experienced anesthesiologist prior to surgery using a standardized technique. Periarticular injection will be administered intraoperatively by the operating surgeon according to a standardized institutional protocol. Apart from the assigned analgesic strategy, all participants will receive standardized anesthesia and postoperative multimodal pain management to minimize confounding factors.

The primary objective of the study is to compare the effectiveness of these three analgesic strategies in controlling postoperative pain after hip surgery in older adults. Secondary objectives include assessment of opioid consumption, time to first mobilization, functional recovery, and patient comfort. Safety outcomes will also be evaluated, with particular attention to adverse events relevant to older adults, including hypotension, bradycardia, excessive sedation, nausea, vomiting, and postoperative delirium.

The results of this study are expected to provide clinically meaningful evidence on whether the PENG block offers advantages over standard periarticular injection and whether combining both techniques yields additional benefit. These findings may inform clinical decision-making and contribute to the optimization of postoperative pain management strategies for older adults undergoing hip surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older
* Scheduled for elective or emergency hip surgery (e.g., hip fracture fixation or hip arthroplasty)
* ASA physical status I-III
* Ability to communicate pain intensity using the NRS scale
* Written informed consent obtained from the patient or legal representative

Exclusion Criteria:

* Patient refusal or inability to provide informed consent
* Allergy, intolerance, or contraindication to any study medication: ropivacaine
* Pre-existing neurological deficit or neuropathy of the affected limb
* Coagulopathy (INR >1.5, platelets <100,000/µL) or current therapeutic anticoagulation that contraindicates regional anesthesia
* Infection at or near the injection site
* Severe hepatic or renal impairment
* History of chronic opioid use (daily opioids >30 days before surgery)
* Cognitive impairment or delirium precluding reliable pain assessment
* BMI > 40 kg/m² (if you want to exclude for technical difficulty)
* Patients receiving another regional nerve block for hip surgery
* Pregnancy or breastfeeding
* Participation in another interventional clinical trial within 30 days

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
otal Opioid Consumption | 0-48 hours after surgery
  Cumulative dose of all opioid analgesics administered in the postoperative period, converted to oral morphine milligram equivalents (MME). Values at 24 and 48 hours will be recorded and compared between groups.

SECONDARY OUTCOMES:
Time to First Rescue Analgesia | Within 48 hours after the end of surgery
  Time (in hours) from the end of the PENG block (completion of local anesthetic injection) to the first administration of rescue analgesia (opioid or non-opioid) given for pain intensity ≥4 on the 0-10 Numerical Rating Scale (NRS). Data will be collected from anesthesia records and postoperative medication charts.
Pain Intensity at Rest (NRS 0-10) | 4 hours after surgery
  Pain intensity at rest assessed using the 0-10 Numerical Rating Scale (0 = no pain, 10 = worst imaginable pain). Mean NRS scores at each time point will be compared between groups.
Pain Intensity at Rest (NRS 0-10) | 8 hours after surgery
  Pain intensity at rest assessed using the 0-10 Numerical Rating Scale (0 = no pain, 10 = worst imaginable pain). Mean NRS scores at each time point will be compared between groups.
Pain Intensity at Rest (NRS 0-10) | 12 hours after surgery
  Pain intensity at rest assessed using the 0-10 Numerical Rating Scale (0 = no pain, 10 = worst imaginable pain). Mean NRS scores at each time point will be compared between groups.
Pain Intensity at Rest (NRS 0-10) | 24 hours after surgery
  Pain intensity at rest assessed using the 0-10 Numerical Rating Scale (0 = no pain, 10 = worst imaginable pain). Mean NRS scores at each time point will be compared between groups.
Pain Intensity at Rest (NRS 0-10) | 48 hours after surgery
  Pain intensity at rest assessed using the 0-10 Numerical Rating Scale (0 = no pain, 10 = worst imaginable pain). Mean NRS scores at each time point will be compared between groups.
Pain Intensity During Movement (NRS 0-10) | 4 hours after surgery
  Pain intensity during standardised hip movement (e.g., flexion or assisted mobilization) assessed using the 0-10 Numerical Rating Scale. Mean NRS scores at each time point will be compared between groups.
Pain Intensity During Movement (NRS 0-10) | 8 hours after surgery
  Pain intensity during standardised hip movement (e.g., flexion or assisted mobilization) assessed using the 0-10 Numerical Rating Scale. Mean NRS scores at each time point will be compared between groups.
Pain Intensity During Movement (NRS 0-10) | 12 hours after surgery
  Pain intensity during standardised hip movement (e.g., flexion or assisted mobilization) assessed using the 0-10 Numerical Rating Scale. Mean NRS scores at each time point will be compared between groups.
Pain Intensity During Movement (NRS 0-10) | 24 hours after surgery
  Pain intensity during standardised hip movement (e.g., flexion or assisted mobilization) assessed using the 0-10 Numerical Rating Scale. Mean NRS scores at each time point will be compared between groups.
Pain Intensity During Movement (NRS 0-10) | 48 hours after surgery
  Pain intensity during standardised hip movement (e.g., flexion or assisted mobilization) assessed using the 0-10 Numerical Rating Scale. Mean NRS scores at each time point will be compared between groups.
Incidence of Postoperative Nausea and Vomiting (PONV) | 0-48 hours after surgery
  Presence of nausea and/or vomiting requiring antiemetic therapy. The proportion of patients with at least one episode of PONV will be recorded and compared between groups
Block-Related Adverse Events, Including Neurological Complications | From block placement until hospital discharge, up to 30 days
  Incidence of complications potentially related to the PENG block or perineural adjuvants, including signs of local anesthetic systemic toxicity, prolonged motor or sensory deficit, nerve injury (evaluated in the postoperative clinic or outpatient nerve injury clinic if required), infection at the injection site, hematoma, or persistent weakness.
Motor Function Preservation (Quadriceps Strength, MRC Scale) | 4 hours after surgery
  Quadriceps muscle strength will be evaluated using the Medical Research Council (MRC) scale, ranging from 0 (no contraction) to 5 (normal power), at 4, 8, 12, 24, and 48 hours to detect any motor impairment associated with the applied regional anesthesia
Motor Function Preservation (Quadriceps Strength, MRC Scale) | 8 hours after surgery
  Quadriceps muscle strength will be evaluated using the Medical Research Council (MRC) scale, ranging from 0 (no contraction) to 5 (normal power), at 4, 8, 12, 24, and 48 hours to detect any motor impairment associated with the applied regional anesthesia
Motor Function Preservation (Quadriceps Strength, MRC Scale) | 12 hours after surgery
  Quadriceps muscle strength will be evaluated using the Medical Research Council (MRC) scale, ranging from 0 (no contraction) to 5 (normal power), at 4, 8, 12, 24, and 48 hours to detect any motor impairment associated with the applied regional anesthesia
Motor Function Preservation (Quadriceps Strength, MRC Scale) | 24 hours after surgery
  Quadriceps muscle strength will be evaluated using the Medical Research Council (MRC) scale, ranging from 0 (no contraction) to 5 (normal power), at 4, 8, 12, 24, and 48 hours to detect any motor impairment associated with the applied regional anesthesia
Motor Function Preservation (Quadriceps Strength, MRC Scale) | 48 hours after surgery
  Quadriceps muscle strength will be evaluated using the Medical Research Council (MRC) scale, ranging from 0 (no contraction) to 5 (normal power), at 4, 8, 12, 24, and 48 hours to detect any motor impairment associated with the applied regional anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Reysner, MD PhD, Study Chair — Poznan University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in publications arising from this study will be made available to qualified researchers upon reasonable request. Shared data will include baseline characteristics, outcome measures, and safety data necessary to reproduce the main analyses. All data will be fully anonymized prior to sharing to protect participant privacy.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available beginning 6 months after publication of the primary results and will remain available for 5 years following publication.
Access Criteria: Access to the data will be granted to researchers who provide a methodologically sound research proposal. Requests must be approved by the principal investigator and the local ethics committee, if required. Data will be shared under a data use agreement and may be used only for non-commercial scientific research purposes.